CLINICAL TRIAL: NCT02301689
Title: SchlaHF-XF- Register. Sleep Disordered Breathing in Heart Failure Register
Brief Title: SchlaHF-XT-Register. Sleep Disordered Breathing in Heart Failure Register
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: MA120814
Record Dates: First submitted 2014-09-17; First posted 2014-11-26 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure (HF)
Keywords: Heart failure; Chronic heart failure; Sleep disordered breathing; Sleep apnea; Positive Airway Pressure
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure patients

SUMMARY:
The SchlaHF XT Registry is a longitudinal study of patients with heart failure (HF). The study aims to understand the importance of diagnosis and treatment of sleep disordered breathing (SDB) on HF with the following questions:

How often does SDB occur in HF? What forms of SDB occur and how are they treated? How does SDB develop over time? How does the heart failure therapy affect SDB? What is the treatment adherence of patients treated? Does SBD and its treatment affect the survival of heart failure patients?

ELIGIBILITY:
Inclusion Criteria:

* diagnose chronic heart failure, at least 3 months prior to diagnosis
* Age 18 years
* Signed informed consent

Exclusion Criteria:

* Existing Positive Airway Pressure (PAP) therapy or long-term oxygen therapy
* Lack of capacity to consent
* minors
* persons who are housed on judicial or administrative order in an institution
* pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients with Heart failure (HF). HF is defined as a symptom complex of shortness of breath and rapid fatigability on the basis of cardiac disease (World Health Organisation).
Sampling Method: Probability Sample
Enrollment: 4749 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Number of heart failure patients with sleep disordered breathing (apnea hypopnoea index >5) | 5 years
  Assess the changes in prevalence of SDB in HF from baseline to 5 years

SECONDARY OUTCOMES:
Number of heart failure patients with sleep disordered breathing (apnea hypopnea index >5) when exposed to sleep disordered breathing treatment | 5 years
  Assess changes in sleep disordered breathing when exposed to treatment from baseline to 5 years
Number of heart failure patients with sleep disordered breathing (apnea hypopnea index >5) when exposed to Heart Failure treatment | 5 years
  Assess changes in SDB when the patient is treated with heart failure therapy
Number of patients adherent to sleep disordered breathing treatment as measured by device reported usage hours | 5 years
  Assess adherence rates to treatment
Number of deaths of patients with HF and sleep disordered breathing (apnea hypopnoea index >5) who are treated for sleep disordered breathing | 5 years
  Assess survival rates of HF patients who are treated for sleep disordered breathing

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Oldenburg, MD, Principal Investigator — Heart and Diabetes Centre NRW
Locations (1):
- Heart and Diabetes Centre, Bad Oeynhausen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Arzt M, Oldenburg O, Graml A, Schnepf J, Erdmann E, Teschler H, Schoebel C, Woehrle H; SchlaHF-XT investigators. Prevalence and predictors of sleep-disordered breathing in chronic heart failure: the SchlaHF-XT registry. ESC Heart Fail. 2022 Dec;9(6):4100-4111. doi: 10.1002/ehf2.14027. Epub 2022 Sep 2. PMID 36052740